CLINICAL TRIAL: NCT04693338
Title: Assessing the Usability and Workflow Impact of a Mobile-Based Breast Cancer Survivorship Care Plan in the Oncology Practice
Brief Title: Interactive Care Plan for the Monitoring of Symptoms and Recovery in Patients With Stage 0-III Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-002448; NCI-2020-07744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-002448 (Other: Mayo Clinic in Rochester); P30CA015083 (NIH)
Record Dates: First submitted 2020-10-12; First posted 2021-01-05 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (ICP) (Experimental): Patients complete surveys for 4 common symptoms: fatigue, hot flashes, insomnia, and sexual dysfunction and receive educational material via mobile app to help with bothersome symptoms. Patients also complete questionnaires.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Supportive Care

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive ICP tasks
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This phase I trial evaluates how well a mobile device-based breast cancer survivorship interactive care plan works in monitoring symptoms and recovery in patients with stage 0-III breast cancer. The interactive care plan provides patients with individualized, 'just in time' education materials to promote self-management for those reporting difficult to control symptoms, as well as escalations to contact their care team for signs or symptoms concerning for cancer coming back (recurrence). The interactive care plan may help alleviate the symptoms of fatigue, insomnia, hot flashes, and sexual dysfunction; increase physical activity level and improve quality of life in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility and usability of the breast cancer (BC) survivorship interactive care plan (ICP) as designed.

II. To determine the behavioral, toxicity symptom burden and quality of life (QOL) changes in patients engaged with the ICP.

III. To assess clinical workflow impact by the introduction of the ICP in the BC survivor practice.

OUTLINE:

Patients complete surveys for 4 common symptoms: fatigue, hot flashes, insomnia, and sexual dysfunction and receive educational material via mobile application (app) to help with bothersome symptoms. Patients also complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed and treated for breast cancer -- having a biopsy-proven, stage 0-III breast cancer and are within 12 months of completion of loco-regional breast cancer treatment and (as indicated) neoadjuvant and/or adjuvant chemotherapy. Ongoing treatment with adjuvant endocrine, bisphosphonate, and single-agent, HER2-directed therapy during the study period is allowed
* Willing to install an application (APP) on personal smart device

Exclusion Criteria:

* Unwilling to return to Mayo Clinic for routine follow-up visits
* Unwilling to use the Mayo Clinic Mobile App
* Unable to provide consent
* Unable to speak or read English
* Unable to participate in mild activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Symptoms assessment response rate | 12 months
  Will assess the total response rate of all surveys administered over the course of the study. The interaction with the educational materials and reminders will be similarly assessed as a total proportion of interaction with the materials and reminders.

SECONDARY OUTCOMES:
Change in patient behavior (activity) | Baseline up to 12 months
  Will be assessed, using McNemar's test to detect any differences.
Change in toxicity symptom burden | Baseline up to 12 months
  Will be assessed using a paired t-test.
Change in quality of life (QOL) | Baseline up to 12 months
  The statistical significance of this outcome will be tested using a paired t-test to compare baseline and study end QOL questionnaire completion
Clinical workflow impact measured by implementation of the breast cancer survivorship interactive care plan in the practice | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniela L Stan, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT04693338/ICF_000.pdf